CLINICAL TRIAL: NCT06687356
Title: Study on the Application of Intraoperative Optical Coherence Tomography Technique in the Diagnosis and Treatment of Lens Diseases
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-0993
Record Dates: First submitted 2024-11-08; First posted 2024-11-13 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Lens Diseases
MeSH Terms: conditions — Lens Diseases | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Traditional surgery (Active Comparator): Without using the intraoperative optical coherence tomography technique during surgery.
  Interventions: Procedure: Conventional surgery
- Surgery with intraoperative optical coherence tomography technique (Experimental): Applying the intraoperative optical coherence tomography technique during surgery.
  Interventions: Procedure: Surgery with Intraoperative Optical Coherence Tomography application

INTERVENTIONS:
Procedure: Surgery with Intraoperative Optical Coherence Tomography application — Surgery with the application of intraoperative optical coherence tomography technique. Intraoperative optical coherence tomography technique can provide intraocular images and show changes in intraocular structures, assisting in analyzing the correlation between preoperative, intraoperative anterior segment structural changes and postoperative surgical effects in patients with lens diseases.
  Other Names: Surgery with Intraoperative OCT application
  Arms: Surgery with intraoperative optical coherence tomography technique
Procedure: Conventional surgery — Conventional lens surgery, without the application of intraoperative optical coherence tomography technique.
  Arms: Traditional surgery

SUMMARY:
Accurately assessing and dealing with anterior segment changes in the eyes of patients with lens diseases can better guide the operation details during surgery and make reasonable plans for possible intraoperative and postoperative complications. Applying the intraoperative optical coherence tomography technique, this study analyzes the correlation between preoperative, intraoperative anterior segment structural changes and postoperative surgical effects in patients with lens diseases, and evaluates the clinical benefits of intraoperative optical coherence tomography technique in lens surgery. This study is intended to further improve the diagnosis and treatment quality of clinical lens diseases.

DETAILED DESCRIPTION:
In the eyes of patients with lens diseases, there are often some special anterior segment changes, including ectopia lentis, abnormal lens morphology, and rupture of the lens capsule. These changes can be caused by ocular trauma, congenital anomalies, or be secondary to other ocular diseases and systemic diseases. Accurately assessing and dealing with these anterior segment changes can better guide the operation details during surgery and make reasonable plans for possible intraoperative and postoperative complications. This study is based on intraoperative optical coherence tomography technique, analyzes the correlation between preoperative, intraoperative anterior segment structural changes and postoperative surgical effects in patients with lens diseases, and evaluates the clinical benefits of intraoperative optical coherence tomography technique in lens surgery. This study is intended to further improve the diagnosis and treatment quality of clinical lens diseases.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged over 18 years old, with lens opacity or abnormal position, and other conditions meeting the surgical indications, needing lens surgery treatment, with or without anterior segment structural changes.

Exclusion Criteria:

* Combined with other eye diseases that seriously affect visual prognosis, serious systemic diseases and other conventional contraindications for lens surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2024-11-27 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Successful implantation rate of intraocular lens | through study completion, an average of 1 year
  Implantation rate of intraocular lens after surgery.
Intraocular lens position after implantation | 1day, 1 week and 1 month postoperation
  The location of intraocular lens after surgery, observed through slit - lamp and anterior segment optical coherence tomography.

SECONDARY OUTCOMES:
Postoperative corneal incision closure status | 1day, 1 week postoperation
  Corneal incision closure status after surgery, observed through slit - lamp and anterior segment optical coherence tomography.
Visual function | 1day, 1 week, 1 month, 3month postoperation
  Best corrected visual acuity (BCVA) measured using a decimal chart Best corrected visual acuity (BCVA) measured using a decimal chart

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China